CLINICAL TRIAL: NCT07129642
Title: The Efficacy and Safety of Allogenic Anti-CD19 CAR-T Cell Therapy for Refractory Graves' Disease
Brief Title: Allogeneic Anti-CD19 CAR-T for Refractory Graves' Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xiaoying Li, Professor, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-217R
Record Dates: First submitted 2025-08-06; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Graves Disease
Keywords: CAR-T; refractory Graves disease; TSH receptor antibody
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental)
  Interventions: Biological: Allogeneic CAR-T

INTERVENTIONS:
Biological: Allogeneic CAR-T — The participants will receive one dose of allogeneic CAR-T

SUMMARY:
Graves' disease is an autoimmune disease. The TSH receptor antibody(TRab) produced by B cells drives the production of thyroid hormone, which causes systemic disorders and thyroid eye disease. The purpose of this study is to investigate the efficacy and safety of allogeneic anti-CD19 CAR-T for refractory Graves' disease.

The participants with refractory Graves' disease will receive a single dose of allogeneic anti-CD19 CAR-T and be regularly seen for the change of serum TRab, FT3, FT4 and clinical presentations, as well as any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with refractory Graves disease, which is defined as meeting any one of the following criteria: a. Failure to discontinue medication after continuous standard antithyroid therapy for ≥ 3 years; b. Hyperthyroid state requiring medication after receiving ≥ 2 times of radioiodine therapy (with the last dose of radioiodine administered at least 6 months prior); c. Relapse ≥ 2 times after cessation of medication upon meeting the criteria for treatment discontinuation.
* Serum TRAb ≥ 3 times greater than normal range (≥ 5 IU/L)
* Positive expression of CD19 on peripheral blood B cells determined by flow cytometry.
* Participation in this clinical study is willing to sign an informed consent with good compliance with treatment and follow-up.

(Criteria for treatment discontinuation is define as receiving continuous anti-thyroid drug therapy for ≥18 months, and maintaining euthyroid status for ≥6 months, plus negative TRAb and TSI. Relapse is defined as recurrence of hyperthyroidism and positive TRAb/TSI after meeting the criteria for treatment discontinuation and stopping medication.)

Exclusion Criteria:

* History of severe drug allergies or allergic constitution;
* Presence or suspicion of uncontrolled infections requiring intravenous treatment (fungal, bacterial, viral or other);
* Presence of central nervous system disorders (including epilepsy, psychosis, cerebrovascular accident, encephalitis, CNS vasculitis, etc);
* Presence of clinically significant heart diseases (e.g., angina pectoris, myocardial infarction, heart failure, severe arrhythmias, etc);
* Subjects with congenital immunoglobulin deficiency;
* Patients with malignant tumors;
* Subjects who are: 1. HBsAg or HBcAb positive with detectable peripheral blood HBV DNA; 2. HCV antibody positive with detectable HCV RNA; 3. Positive HIV antibody; 4. Syphilis test positive;
* Subjects with psychiatric disorders or severe cognitive dysfunction;
* Hematopoietic function: a. White blood cell count < 3.5×10^9/L b. Neutrophil count < 1.5 x 10^9/L; c. Hemoglobin < 110g/L.
* Liver function: ALT> 3×ULN, AST > 3×ULN, TBIL > 2.5×ULN.
* Renal function: creatinine clearance rate (CrCl) < 60 ml/minute (calculated based on Cockcroft/Fault formula).
* Cardiac function: LVEF < 55%
* Coagulation function: International standardized ratio (INR) ≥ 1.5×ULN, prothrombin time(PT) >1.5 × ULN.
* Participation in other clinical trials within 3 months prior to enrollment;
* Pregnancy or planning pregnancy;
* Other conditions considered by investigators as unsuitable for participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Remission of Graves disease | From baseline to 12 months after infusion of CAR-T cells
  Sustained euthyroid status without anti-thyroid medication for ≥3 months
Incidence of Adverse Events | From baseline to 6 months after infusion of CAR-T cells
  Assessed using the CTCAE v5.0 standards

SECONDARY OUTCOMES:
Anti-Thyrotropin receptor antibody (TRAb) | From baseline to 12 months after infusion of CAR-T cells
  Serum TRAb titers at 6 months and 12 months after infusion of CAR-T cells
Thyroid stimulating immunoglobulin (TSI) | From baseline to 12 months after infusion of CAR-T cells
  Serum TSI titers at 6 months and 12 months after infusion of CAR-T cells
thyroid peroxidase antibody (TPOAb) | From baseline to 12 months after infusion of CAR-T cells
  Serum TPOAb titers at 6 months and 12 months after infusion of CAR-T cells
Thyroglobulin antibody (TgAb) | From baseline to 12 months after infusion of CAR-T cells
  Serum TgAb titers at 6 months and 12 months after infusion of CAR-T cells
Thyroid volume | From baseline to 12 months after infusion of CAR-T cells
  Size of thyroid measured and calculated by ultrasound at 6 months and 12 months after infusion of CAR-T cells
PK parameters - CAR gene copy number | From baseline to 3 months after infusion of CAR-T cells
  Dynamic change in the CAR gene copy number in peripheral blood after infusion of CAR-T cells
PK parameters - CAR-T cell count | From baseline to 3 months after infusion of CAR-T cells
  Dynamic change of CAR-T cell count in peripheral blood after infusion of CAR-T cells

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying LI, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: After publication.
Access Criteria: IPD and supporting information will be avaible to researchers upon reasonable request (e.g. with a practical and meaningful research proposal).